CLINICAL TRIAL: NCT06535113
Title: Decoding the Inflammasome Influence on Treatment Response in Acute Myeloid Leukemia
Acronym: Inflamm-AML
Status: Recruiting | Type: Observational
Sponsor: Ciceri Fabio (Other)
Collaborators: Azienda Ospedaliera Bianchi-Melacrino-Morelli (Other)
Responsible Party: Sponsor-Investigator, Ciceri Fabio, Prof. MD Director, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: PNRR-MCNT1-2023-12377456
Record Dates: First submitted 2024-07-29; First posted 2024-08-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Leukemia; Chemotherapy; inflammation; transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — bone marrow, biopsies, and peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- acute myeloid leukemia (AML) patients treated in the clinical units: acute myeloid leukemia (AML) patients treated in the clinical units
  Interventions: Other: Clinical Practice

INTERVENTIONS:
Other: Clinical Practice — All the procedures in Study will be conducted as per Clinical practice for the pathology and all the samples will be collected according to ELN guidelines.
  There are no additional procedures but will be additionally collected up 20ml of peripheral blood and up to 15ml of Bone Marrow Aspirate at the same time of clinically indicated diagnostic procedures.

SUMMARY:
The study is designed as a collection of biological samples of newly diagnosed acute myeloid leukemia (AML) patients treated in the clinical units involved. Samples of peripheral blood (PB) and bone marrow (BM) will be analyzed to determine the Inflammasome profile before and after a first-line chemotherapy treatment.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a highly aggressive and unfavorable malignancy primarily affecting bone marrow (BM) myeloid cells, particularly in older individuals. The standard treatment for fit, intermediate and high-risk patients involves chemotherapy followed by allogeneic hematopoietic stem cell transplantation (HSCT). However, around 60% of patients experience relapse, requiring second-line therapies that offer a reduced likelihood of achieving a permanent cure.

Inflammation significantly influences AML development, progression, leukemic cell behavior, and treatment response. Interactions between leukemic cells and microenvironment promote their growth, survival, and drug resistance. The inflammasome, an intracellular complex crucial for promoting inflammation, triggers the release of the proinflammatory cytokines interleukin (IL)-1beta and IL-18, and induces pyroptosis (inflammatory cell death) in response to inflammatory stimuli. There is growing evidence suggesting a link between the inflammasome and AML, with components of the inflammasome being overexpressed in leukemic cells. The precise mechanisms by which the inflammasome and its activation pathways influence AML still need to be fully understood.

We speculate that excessive inflammasome activity in AML disrupts the balance of cytokine production, leading to chronic inflammation, which interferes with the normal development and function of hematopoietic cells in the BM microenvironment. This heightened inflammasome signature could impact the way patients respond to chemotherapy, potentially altering inflammatory processes, ultimately reducing the efficacy of the treatment. Variations in inflammasome activation among AML patients may explain differences in treatment outcomes, including response rates, hematopoietic recovery, remission duration, and overall survival.

Understanding the molecular mechanisms involved in AML, particularly the role of the inflammasome, could allow a better disease risk stratification and the development of potential targeted therapies and interventions, which could improve treatment outcomes. More specifically, identifying potential therapeutic targets within the inflammasome pathway, may drive to the design of new treatment strategies, precisely aimed at correcting inflammasome dysregulation in AML. From the clinical point of view, these insights could assist healthcare professionals in taking informed decisions in the management of AML patients. By modulating inflammasome activity or targeting specific pathway components, we could develop personalized treatment approaches tailored to individual patient needs, optimizing treatment response and possibly minimizing chemotherapy-related side effects. This personalized approach has the potential to enhance the quality of life for patients, reduce complications, and increase the overall effectiveness of treatments.

During the Study period patients referring to the clinical centers will undergo the standard diagnostic and therapeutic process for their pathology, according to international guidelines. For all the patients that will agree to participate, clinical data and biological samples will be analyzed for the aims of the Study. The retrospective part of the data and material collection must have bio-banked material in compliance with the ethics and regulatory standards for the research purpose.

Due to the Observational nature of the Study, all diagnostic procedures and treatments applied are considered common practice. All treatments comply with the ATC Code L01, the different schemes of treatment could be categorized under an "intensive" or "non intensive" protocol.

Commonly used intensive induction regimens are:

* 3+7; = daunorubicine 60 mg/m^2 day 1-3 + cytarabine as continue IV infusion 100/200 mg/m^2 day 1-7
* 3+7; + midostaurine 50 mg every 12 hours, day 8-21
* 3+7; + gemtuzumab ozogamicin 3 mg/m^2 day 1, 4, 7
* CPX-351 (daunorubicin 44 mg/cytarabine 100 mg) IV days 1, 3, 5 Commonly used intensive consolidation schemes include intermediate/high dose cytarabine or CPX-351. Midostaurine, gemtuzumab ozogamicin, daunorubicine may be added as per guidelines.

Non intensive induction and consolidation schemes include: azaticidine (75 mg/m^2) day 1-7 + Venetoclax at variable dose.

For the retrospective collection of samples, the preceding version of ELN guidelines (2017) will be appliedThe main hypothesis of the study is that an excessive inflammasome activity in AML disrupts the balance of cytokine production, leading to a clinically relevant inflammatory state, which interferes with the response to chemotherapy.

In two years, we plan to recruit 80 adult participants with a new diagnosis of AML undergoing first line chemotherapy treatment.

The protocol is a multicenter, national, observational study; indeed, it is based on the Clinical Practice and is aimed at gathering information from the biological samples collected during the diagnosis process and after a first line treatment. The Study will be prospective and retrospective. The total duration of enrolment will be from August 2024 to January 2026, the observation period will be up to 6 months. The information about the treatment and the assessment on disease response/relapse/progression will be collected for stratification and monitoring purpose. Retrospectively, specimens, demographical and clinical information are retrieved from AML patients previously recruited by UO1 will be utilized. Prospectively, new AML patients will be recruited. UO1 recruits AML patients, collects biological samples at diagnosis and after chemotherapy, processes, and biobanks specimens, and conducts functional inflammasome assays, gene expression analysis, and immunophenotyping of AML blasts in peripheral blood and bone marrow. Additionally, immunohistochemistry is performed on bone marrow biopsies. UO2 recruits AML patients, processes and cryobank specimens, and ships samples to UO1. It also produce all diagnostic data for clinical standard of AML blasts in peripheral blood and bone marrow, with immunohistochemistry conducted on bone marrow biopsies.

The biological samples collected for the study include bone marrow, biopsies, and peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Any gender,
* Adults (>18 years old),
* New suspect diagnosis of acute myeloid leukemia (ELN2022 Criteria)
* Capable of comprehend the study and the consent form,
* Willing to sign the informed consent for the study.

For the retrospective population we will select:

biological samples (BM Biopsies, BM Aspirates and PB) already banked upon research purpose informed consent and collected from the 01/06/2006 up to 01/06/2024 from adults patients with diagnosis of acute myeloid leukemia according to ELN2017 Criteria.

Exclusion Criteria:

* Pediatric patients (<18 years old),
* Patients unable or unwilling to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on the population seen at the clinical centers as per common practice. The subjects eligible will be identified during the clinical practice diagnostic process for AML.
  The study will involve a total of 80 subjects based on the statistical design for the Study. The Coordinating Unit of the Study will include at least 55 subjects, the Other cooperating Centers will provide the remaining subjects.
  The retrospective samples will be identified through Biobanking Records in the pool of samples stocked and we estimate around 25% of the total population included (~20 subjects).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Inflammasome Activity | At diagnosis, in case of treatment failure and at 6 months after first line chemotherapy initiation
  The outcome variable is the inflammasome activation in AML blasts (PB e BM)

SECONDARY OUTCOMES:
Correlation Inflammasome and Therapy | At diagnosis, in case of treatment failure and at 6 months after first line chemotherapy initiation
  To evaluate the correlation between inflammasome activity and response to chemotherapy in patients with AML

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - GOM Bianchi Melacrino Morelli, Reggio Calabria, Calabria
  - IRCCS Ospedale San Raffaele, Milan, Milan

IPD SHARING:
Plan to Share IPD: No
all Data that underlie results will be published on a peer reviewed paper as for legal requirments